CLINICAL TRIAL: NCT03902886
Title: Biomechanics and Motor Control of the First 6 Months of Independent Walking for Children With Unilateral Cerebral Palsy
Brief Title: Independent Walking Onset of Children With Cerebral Palsy
Acronym: BB-AQM
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: BB-AQM ( 29BRC18.071)
Record Dates: First submitted 2018-10-22; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2018-10

CONDITIONS: Cerebral Palsy
Keywords: toddlers, gait
MeSH Terms: conditions — Cerebral Palsy | interventions — Gait Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cerebral palsy infants: gait analysis
  Interventions: Diagnostic Test: gait analysis
- typically developed infants: gait analysis
  Interventions: Diagnostic Test: gait analysis

INTERVENTIONS:
Diagnostic Test: gait analysis — gait analysis using an optoelectronic system and a surface EMG

SUMMARY:
This study will focus the gait analysis, using an optoelectronic system, of children with unilateral cerebral palsy compared to typically developed children in the first 6 months of independent walking.

ELIGIBILITY:
Inclusion Criteria:

* Maximum age of 3 years old
* Independent walking experience of maximum 6 months
* Ability to walk 5 m without falling or needing a technical assistance
* A right or left hemiplegia in a predictive clinical context of a CP at the age of 2 years

Exclusion Criteria:

* History of lower limb musculoskeletal trauma in the last 6 months
* A known skin allergy to any adhesive product
* History of lower limb musculoskeletal surgery
* History of BTX injections into the lower limbs muscles in the last 3 months

Max Age: 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 10 toddlers with unilateral CP will be compared to 10 toddlers typically developed. The populations will have maximum 6 months of walking experience.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

PRIMARY OUTCOMES:
The lower limbs Global Profile Score during gait | All the data collection and analysis wil be done within 2 months from the start point of the study.
  Data will be collected from gait analysis of unilateral CP children and the Global Profile Score, characterizing the overall kinematics of the pelvis and lower limbs, during gait, will be compared those of a typical developed children group matched in walking experience. Mann Whitney U test will be used for this comparison.

CONTACTS AND LOCATIONS:
Locations (2):
- CHRU de Brest, Brest, France
- Centrul National Clinic Recuperare Copii "Dr. N. Robanescu", Bucharest, Romania